CLINICAL TRIAL: NCT03445351
Title: Effect of Exercise on Quality of Life, Sleep, and Biomarkers in People With HIV/AIDS
Brief Title: Quality of Life, Sleep, and Biomarkers in People With HIV/AIDS
Acronym: PLHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JULIANY DE SOUZA ARAUJO (Other)
Responsible Party: Sponsor-Investigator, JULIANY DE SOUZA ARAUJO, CLINICAL TEACHER, Universidade Federal do Rio Grande do Norte
Organization: Universidade Federal do Rio Grande do Norte (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AFISA
Record Dates: First submitted 2017-11-21; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: HIV/AIDS and Infections; Disorder Sleep; Lipodystrophy
Keywords: Exercise Therapy;; Sleep;; ; Immune Markers;; HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Parasomnias; Lipodystrophy

STUDY DESIGN:
Intervention Model Description: Intervention study, prospective, a cohort with 17 PLHA participants of the exercise program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic, resistance and concorrent (Experimental): The group underwent exercise program with protocols of resistance training, aerobic training and concurrent training, with frequency of three times per week.
  Interventions: Other: Aerobic, resistance and concorrent.

INTERVENTIONS:
Other: Aerobic, resistance and concorrent. — All protocols followed the American College of Sports Medicine (ACSM) guidelines , with frequency of three times per week, duration between 40-50 minutes, low to high intensity, modified according to the physical needs of each participant, respecting the physical training principles.

SUMMARY:
Aim: Evaluate the influence of exercise, in different times, on quality of life, sleep and clinical parameters in people living with HIV/AIDS (PLHA). Methods: Intervention study, prospective.

DETAILED DESCRIPTION:
Aim: Evaluate the influence of exercise, in different times, on quality of life, sleep and clinical parameters in people living with HIV/AIDS (PLHA). Methods: Intervention study, prospective, a cohort with 17 PLHA participants of the exercise program, higher than 18 years, under antiretroviral therapy with CD4+ ≥ 350/mm3. Research Ethical Committee of the institution approved the study and the participants sign the informed consent and informed. All subjects underwent an exercise program in conformity to American College of Sports Medicine, 3 times per week during 40 minutes. Were evaluated the quality of life (QoL) with the Quality of Life - HAT - QoL and the sleep quality (SQ) with the Pittsburg questionnaire. The subjects were evaluated before the start of exercise program and in three times: short-term (2 to 4 months), medium-term (between 5 and 17 months) and long-term (between 18 to 25 months).

ELIGIBILITY:
Inclusion Criteria:

* Must have age ≥ 18 years old;
* diagnosis of HIV/AIDS;
* use of antiretroviral therapy;
* Must have lymphocyte T CD4+ cell count ≥ 350 cel/mm3
* Must have physical fitness by the assistant physician.

Exclusion Criteria:

* pregnancy;
* severe hearing deficiency.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2013-01-20 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2016-09-13 (Actual)

PRIMARY OUTCOMES:
Quality of life | 24 MONTHS
  A translation adapted and validated for Brazil of the HIV/AIDS Targeted Quality of Life questionnaire (HAT-QoL) developed by Holmes & Shea, was used . The HAT-QoL present 34 questions divided in nine domains: Overall Function (OVEFUN), Life Satisfaction (LISA), Health Worries (HEAWOR), Financial Worries (FINWOR), Medication Concerns (MEDCON), HIV Mastery (HIVMAS), Disclosure Worries (DISWOR), Provider Trust (PROTRU) and Sexual Function (SEXFUN). The score ranges from 0 to 100. The responses have a five-point Likert scale: "all the time", "most of the time", "part of the time", "little time" and "never". In each domain, zero is the lowest score and 100 the best score possible. The higher the score, the lower the impact of HIV infection on the individuals' quality of life.

SECONDARY OUTCOMES:
Quality of sleep | 24 MONTHS
  For the QoS the Pittsburgh Sleep Quality Index validated for Brazilian population, was applied. This scale is composed of 19 items that evaluate aspects related to sleep latency, duration, usual efficiency, sleep disturbance, use of hypnotic drugs and daytime dysfunction in the last month. Scores smaller than 5 define good sleep quality; values ranging between 6 to 11 bad sleep quality and values greater than 11 sleep disturbance. To answer the questionnaires, the subjects were oriented to think about the QoL and QoS in the previous four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: RAFAELA MEDEIROS, Principal Investigator — Universidade Federal do Rio Grande do Norte

IPD SHARING:
Plan to Share IPD: No